CLINICAL TRIAL: NCT04285112
Title: SPRINT: Signature for Pain Recovery IN Teens
Acronym: SPRINT
Status: Active, not recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: University of Toronto (Other); The Hospital for Sick Children (Other); University of Barcelona (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Laura E Simons, Professor, Stanford University
Other Study IDs: 2019-1006; 52963 (Other: Stanford)
Record Dates: First submitted 2020-02-23; First posted 2020-02-26 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Pain, Chronic; Pain; Joint Pain; Musculoskeletal Pain
Keywords: Pediatric pain; pain
MeSH Terms: conditions — Chronic Pain; Pain; Arthralgia; Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To identify biological and phenotypic prognostic markers of recovery vs. persistence of pain and functional disability in adolescents with chronic musculoskeletal pain.

DETAILED DESCRIPTION:
Up to 5% of adolescents (~3.5 million in the US alone) suffer from high impact chronic musculoskeletal (MSK) pain, affecting all life domains and posing a significant economic burden. Current treatments for chronic MSK pain are suboptimal and have been tied to the opioid crisis. Only ~50% of adolescents with chronic MSK pain who present for multidisciplinary pain treatment recover, as measured by clinical endpoints of pain severity and functional disability. Discovery of robust markers of the recovery vs. persistence of pain and disability is essential to develop more resourceful and patient-specific treatment strategies and to conceive novel approaches that benefit patients who are refractory. Given that chronic pain is a biopsychosocial process, the discovery and validation of a prognostic and robust signature for pain recovery vs. persistence requires measurements across multiple dimensions in the same patient cohort in combination with a suitable 'big data' computational analysis pipeline for the extraction of reliable and cross-validated results from a multilayered and complex dataset. The research team is well positioned to execute the study aims with: (1) A highly skilled and experienced team of scientists and clinicians from Stanford University, University of Toronto/Hospital for Sick Children, and Cincinnati Children's Hospital Medical Center; (2) A standardized specimen collection, processing, storage, and distribution system, leveraging Stanford Biobank's platform, BioCatalyst, to aggregate the sample inventory with clinical annotations for an accessible, virtual biobank, within the Signature of Pain Recovery IN Teens (SPRINT) Biobank and Analysis Core (SBAC); (3) Cutting-edge preliminary data implicating novel candidates for neuroimaging, immune, quantitative sensory, and psychological markers for discovery; and (4) Expertise in machine learning approaches to extract reliable and prognostic bio-signatures from a large and complex data set. The research team expects that the results from this project will facilitate risk stratification in patients with chronic MSK, a more resourceful selection of patients who are likely to respond for undergoing current multidisciplinary pain treatment approaches, and new insight into biological and behavioral processes that may be exploited to develop novel strategies profiting those who are refractory.

For the R61/Discovery Phase Aim individuals will be thoroughly characterized via biological (i.e. brain structure and function, immune, sensory profiles), psychological state, and clinical endpoint (i.e., pain intensity, disability) data. Unbiased machine learning algorithms will identify a multivariate model comprised of the most prognostic biological, psychological, and clinical endpoints. The model will classify adolescents with and without resolving chronic MSK pain after a state-of-the art multidisciplinary pain treatment intervention. R33/Validation Phase Aim will validate the biological signature derived in the R61 study. This signature will be useful for a range of adolescent-based clinical trials in which identification of the highest risk individuals is necessary, providing a clinically actionable intervention algorithm.

ELIGIBILITY:
Inclusion Criteria:

1. The child has a diagnosis of Chronic widespread pain or Chronic primary musculoskeletal pain (other than orofacial) derived from ICD-11 (MG30.0; chronic primary pain is pain in 1 or more anatomic regions that persists for > 3 months, is associated with significant distress or functional disability and cannot be better explained by another chronic pain condition (e.g., arthritis, lupus)
2. Age between 11-18 years
3. Moderate to Severe Functional Disability (FDI ≥13)
4. English proficiency (reading, speaking)
5. Moderate to severe average pain (VAS ≥30/100)

Exclusion Criteria:

1. Significant cognitive impairment (e.g., severe brain injury)
2. Claustrophobia
3. Significant medical disease (e.g., systemic or central nervous system)
4. Severe psychiatric or neurological conditions (e.g., eating disorder, psychosis)
5. Pregnancy
6. MRI incompatibility (braces, pacemaker)
7. Weight > 285 lbs.
8. History of > 1 month opioid treatment.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents with chronic primary musculoskeletal pain
Sampling Method: Non-Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity and Unpleasantness | 3 months after baseline assessment
  Pain Intensity and Unpleasantness on visual analogue scale(VAS). VAS scores range from 0 to 100 with higher scores indicating worse pain.
Functional Disability | 3 months after baseline assessment
  Functional Disability Inventory (FDI) total score. FDI scores range from 0 to 60 with higher scores indicating higher levels of functional disability.

CONTACTS AND LOCATIONS:
Overall Officials: Laura E Simons, PhD, Principal Investigator — Stanford University
Locations (4):
- United States (2):
  - Stanford University, Palo Alto, California
  - Cincinnati Children's Hospital, Cincinnati, Ohio
- Hospital for Sick Children, Toronto, Ontario, Canada
- University of Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Resource sharing plan. Scientific resources produced in the course of this work are valuable for the scientific community. We are committed to open access publication and data sharing. After findings have been published or are submitted for publication, we will upload all data on applicable repositories (https://www.nature.com/sdata/policies/repositories). Potential current repositories include: OpenPain http://www.openpain.org/, OpenNeuro https://openneuro.org/, Open Science Framework https://osf.io/, flowrepository http://flowrepository.org/, ImmPort https://www.immport.org/shared/home.
Time Frame: After findings have been published or are submitted for publication, we will upload all data on applicable repositories.
Access Criteria: Any interested party will need to submit a request to the study team.

REFERENCES:
- [Derived] Simons L, Moayedi M, Coghill RC, Stinson J, Angst MS, Aghaeepour N, Gaudilliere B, King CD, Lopez-Sola M, Hoeppli ME, Biggs E, Ganio E, Williams SE, Goldschneider KR, Campbell F, Ruskin D, Krane EJ, Walker S, Rush G, Heirich M. Signature for Pain Recovery IN Teens (SPRINT): protocol for a multisite prospective signature study in chronic musculoskeletal pain. BMJ Open. 2022 Jun 8;12(6):e061548. doi: 10.1136/bmjopen-2022-061548. PMID 35676017